CLINICAL TRIAL: NCT02209298
Title: Evaluation of the Clinical Outcomes of CoreValve in Degenerative Surgical Aortic Bioprosthesis. A Prospective, Observational Post-market Study.
Brief Title: CoreValve VIVA Study Evaluation of the Clinical Outcomes of CoreValve in Degenerative Surgical Aortic Bioprosthesis.
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: MED-02
Record Dates: First submitted 2014-07-31; First posted 2014-08-05 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CoreValve Transcatheter Valve: Medtronic CoreValve SystemTM is designed to replace the native or surgical bioprosthetic aortic heart valve without open heart surgery and without concomitant surgical removal of the failing valve. The support frame is manufactured by Nitinol, which has multi-level, self-expanding properties and is radiopaque. The bioprosthesis is manufactured by suturing valve leaflets and a skirt from a single layer of porcine pericardium into a tri-leaflet configuration. The bioprosthesis is processed with alpha-amino oleic acid (AOA™), which is a compound derived from oleic acid, a naturally occurring long-chain fatty acid. AOA™ is an antimineralization treatment shown to reduce both early and late valvular calcification.
  Interventions: Device: CoreValve Transcatheter Valve

INTERVENTIONS:
Device: CoreValve Transcatheter Valve — Patients should be accepted for TAVI by a multidisciplinary team. The procedure should use the Medtronic CoreValve SystemTM and point of enrolment is the day of the procedure. The choice of prosthesis size and access route (transfemoral, subclavian or direct aortic access) is to be left to the discretion of the operating team. Equally the intraprocedural details (anaesthetic, imaging etc.) will proceed as per usual practice.

SUMMARY:
This observational study is intended to collect real-world (post-approval use) data regarding the clinical utility and performance of the Medtronic CoreValve® System for Transcatheter Aortic Valve Implantation (TAVI).

DETAILED DESCRIPTION:
To collect real-world (post-approval use) data regarding the clinical utility and performance of the Medtronic CoreValve® System for TAVI in patients with failing surgical aortic bioprosthesis who are at high risk for redo surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years old
* Patient has a symptomatic degeneration of aortic bioprosthesis
* Acceptable candidate for elective treatment with the Medtronic CoreValveTM System (according to the most recent version of the Medtronic CoreValveTM Instructions For Use) and in conformity with the local regulatory and reimbursement context
* Logistical Euroscore > 20% or STS > 10% or presence of comorbidities responsible of contra-indication(s) for redo surgery as assessed by at least one cardiac surgeon or patients in whom heart team has assessed the redo surgery at high risk
* The patient or legal representative has been informed of the nature of the procedure and the study and has consented to participate, and has authorized the collection and release of his/her medical information by signing a consent form ("Patient Informed Consent Form")
* The patient is willing and able to comply with requirements of the study, including the 24 months follow-up
* Patient will receive the CoreValveTM device in a degenerated surgical bioprosthesis

Exclusion Criteria:

* Patients in whom anti-platelet and/or anticoagulant therapy is contraindicated
* Patient in whom heart team considers that risk of TAVI is too high with a particular attention for the risk of coronary occlusion
* Patient with prior endocarditis on failed bioprosthesis
* Patient has other medical illness associated with a limited life expectancy (i.e., less than 1 year)
* Patient with LVEF <20%, cardiogenic shock, or hemodynamic compromise requiring pressors or inotropes or mechanical support devices
* Patient with severe mitral disease associated with severe pulmonary hypertension
* Acute coronary syndrome less than 7 days before intervention
* Currently participating in another investigational drug or device study.
* Patient with significant paravalvular regurgitation
* Patient in whom internal diameter prosthesis is equal to 17 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be screened from symptomatic high risk adult patients candidates for an intervention on degenerative surgical aortic bioprosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular death | 30 days post-index procedure
Lack of significant aortic stenosis or insufficiency | 1 year Follow-up

SECONDARY OUTCOMES:
Safety composite endpoint based on VARC-II endpoint definitions | At 30 days and during follow-up visits
Peri-procedural myocardial infarction, major and minor access site complications, major bleeding, stroke, acute kidney injury stage III, new pacemaker implantation, and post-implantation aortic gradient | At 30 days and during follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Didier Tchetche, Dr., Principal Investigator — Clinique Pasteur Toulouse; Jean-Philippe Verhoye, Prof., Principal Investigator — Centre Hospitalier Universitaire, Rennes; Ran Kornowski, Prof., Principal Investigator — Rabin Medical Center, Tel Aviv
Locations (25):
- France (15):
  - CHU Brest, Brest
  - CHU Clermont, Clermont-Ferrand
  - CHU Mondor, Créteil
  - Clinique Parly 2 Le Chesnay, Le Chesnay
  - CHU Lille, Lille
  - HCL CHU Louis Pradel, Lyon
  - CHU La Timone, Marseille
  - Hopital Jacques Cartier, Massy
  - CHU de Nantes, Nantes
  - CHU La Pitié Salpétrière, Paris
  - CHU Bordeaux, Pessac
  - CHU Rennes, Rennes
  - CHU Rangueil Toulouse, Toulouse
  - Clinique Pasteur, Toulouse
  - Tonkin Clinic, Villeurbanne
- Germany (5):
  - Kerckhoff Klinik, Bad Nauheim
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Sana-Herzzentrum Cottbus, Cottbus
  - Hamburg Eppendorf, Hamburg
  - Herzzentrum Leipzig GmbH Leipzig, Leipzig
- Israel (2):
  - Rabin Medical center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Italy (3):
  - Brescia Hospital, Brescia
  - Policlinico San Donato, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa

REFERENCES:
- [Derived] Kornowski R, Chevalier B, Verhoye JP, Holzhey D, Harnath A, Schӓfer U, Teiger E, Manigold T, Modine T, Souteyrand G, Champagnac D, Oh JK, Li S, Tchetche D; VIVA Investigators. Transcatheter Aortic Valve Implantation for Failed Surgical Aortic Bioprostheses Using a Self-Expanding Device (from the Prospective VIVA Post Market Study). Am J Cardiol. 2021 Apr 1;144:118-124. doi: 10.1016/j.amjcard.2020.12.047. Epub 2020 Dec 28. PMID 33383007
- [Derived] Tchetche D, Chevalier B, Holzhey D, Harnath A, Schafer U, Teiger E, Manigold T, Modine T, Souteyrand G, Champagnac D, Oh JK, Li S, Verhoye JP, Kornowski R; VIVA Investigators. TAVR for Failed Surgical Aortic Bioprostheses Using a Self-Expanding Device: 1-Year Results From the Prospective VIVA Postmarket Study. JACC Cardiovasc Interv. 2019 May 27;12(10):923-932. doi: 10.1016/j.jcin.2019.02.029. PMID 31122349